CLINICAL TRIAL: NCT03644277
Title: HANDS: A Multi-Center Clinical Trial to Evaluate the Effectiveness of Intermittent Hypoxia Therapy in Individuals With Spinal Cord Injury
Brief Title: A Multi-Center Clinical Trial in Individuals With Spinal Cord Injury
Acronym: HANDS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Zev Rymer, Principle Investigator, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00206247
Record Dates: First submitted 2018-03-12; First posted 2018-08-23 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Upon enrollment in the study, participants will be randomly assigned to one of five groups, including: massed practice training with dAIH, massed practice training with Sham dAIH, Rapael glove with dAIH, Rapael glove with Sham dAIH, and no training with dAIH.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Massed practice training with dAIH (Experimental): Seek to address gross upper extremity movements, grip and pinch strength, and coordination.The ultimate goal of the session is to achieve a total of 300 repetitions during training.
  Once fitted with the mask, initial recordings of heart rate, blood pressure, and arterial oxygen saturation (SpO2) will be taken. The sequence of hypoxia will consist of 60- 90 seconds of 9-10% O2 (FiO2 0.09), alternating with 60- 90 seconds of 21% O2 (normoxic air FiO2 0.21). The delivery of hypoxia and normoxic air mixtures will be repeated up to 18 times per session each, for a total of up to 45 minutes, to maintain SpO2 at 80-90%.
  Interventions: Other: Acute Intermitted Hypoxia; Procedure: Massed Practise
- Massed practice training with Sham dAIH (Experimental): Seek to address gross upper extremity movements, grip and pinch strength, and coordination.The ultimate goal of the session is to achieve a total of 300 repetitions during training.
  Once fitted with the mask, initial recordings of heart rate, blood pressure, and arterial oxygen saturation (SpO2) will be taken. The sequence of hypoxia will consist of 60- 90 seconds of 9-10% O2 (FiO2 0.09), alternating with 60- 90 seconds of 21% O2 (normoxic air FiO2 0.21). The delivery of hypoxia and normoxic air mixtures will be repeated up to 18 times per session each, for a total of up to 45 minutes, to maintain SpO2 at 80-90%.
  Interventions: Other: Acute Intermitted Hypoxia; Procedure: Massed Practise
- Rapael glove with dAIH (Experimental): The Rapael Smart Glove is a virtual reality hand exoskeleton rehabilitation device. The tasks selected will address gross movement, hand function, and dexterity. Tasks utilized will include, but are not limited to: fly swat, throwing darts, squeezing an orange, catching a baseball, and floating fish. The number of total repetitions and activity outcomes will be recorded.
  Once fitted with the mask, initial recordings of heart rate, blood pressure, and arterial oxygen saturation (SpO2) will be taken. The sequence of hypoxia will consist of 60- 90 seconds of 9-10% O2 (FiO2 0.09), alternating with 60- 90 seconds of 21% O2 (normoxic air FiO2 0.21). The delivery of hypoxia and normoxic air mixtures will be repeated up to 18 times per session each, for a total of up to 45 minutes, to maintain SpO2 at 80-90%.
  Interventions: Other: Acute Intermitted Hypoxia; Other: Rapael Glove
- Rapael glove with Sham dAIH (Active Comparator): The Rapael Smart Glove is a virtual reality hand exoskeleton rehabilitation device. The tasks selected will address gross movement, hand function, and dexterity. Tasks utilized will include, but are not limited to: fly swat, throwing darts, squeezing an orange, catching a baseball, and floating fish. The number of total repetitions and activity outcomes will be recorded.
  Once fitted with the mask, initial recordings of heart rate, blood pressure, and arterial oxygen saturation (SpO2) will be taken. The sequence of hypoxia will consist of 60- 90 seconds of 9-10% O2 (FiO2 0.09), alternating with 60- 90 seconds of 21% O2 (normoxic air FiO2 0.21). The delivery of hypoxia and normoxic air mixtures will be repeated up to 18 times per session each, for a total of up to 45 minutes, to maintain SpO2 at 80-90%.
  Interventions: Other: Acute Intermitted Hypoxia; Other: Rapael Glove
- No training with dAIH (Placebo Comparator): Once fitted with the mask, initial recordings of heart rate, blood pressure, and arterial oxygen saturation (SpO2) will be taken. The sequence of hypoxia will consist of 60- 90 seconds of 9-10% O2 (FiO2 0.09), alternating with 60- 90 seconds of 21% O2 (normoxic air FiO2 0.21). The delivery of hypoxia and normoxic air mixtures will be repeated up to 18 times per session each, for a total of up to 45 minutes, to maintain SpO2 at 80-90%.
  Hearth rate and pulse oximetry will be continuously monitored throughout, and recording will be taken at each alteration in sequence. Blood pressure will be taken upon completion of the total sequence
  Interventions: Other: Acute Intermitted Hypoxia

INTERVENTIONS:
Other: Acute Intermitted Hypoxia — Subjects will be fitted with a latex-free full non-rebreather mask with a custom neoprene head strap, mask and oxygen delivery system are commonly used for altitude training. The mask will first provide a normoxic air (room air) mixture (FiO2 = 0.21) via the mask.
  Other Names: dAIG
Procedure: Massed Practise — Address gross upper extremity movements, grip and pinch strength, and coordination.
  Tasks utilized may include, but are not limited to: lifting a weighted can, squeezing, cutting paper, popping bubble wrap, translating different resistance clothespins, etc. The ultimate goal of the session is to achieve a total of 300 repetitions during training. Task difficulty may be progressed (making it more difficult), if the participant is able to achieve >100 repetitions in less than 15 minutes, on two different occasions. A task may be made easier if the participant is unable to achieve 50 repetitions of a task within 15minutes. Progressing a task may include: changing the task, addition of resistance, increasing the range of motion required for a task to be deemed successful, increasing/decreasing the size of the object used. The number of total repetitions and any item progressions will be recorded.
  Arms: Massed practice training with Sham dAIH; Massed practice training with dAIH
Other: Rapael Glove — The Rapael Smart Glove is a virtual reality hand exoskeleton rehabilitation device. The tasks selected will address gross movement and hand function during a 45 minute session. Additional time may be required for device set up and activity selection/modification. Tasks utilized will include, but are not limited to: fly swat, throwing darts, squeezing an orange, catching a baseball, and floating fish. Tasks will be modified based on participants' perceived fatigue and challenge levels, as determined by a rating from 0-10. The participant goal will be to maintain the task difficulty between a 5-8/10 range. This would depict a moderate to difficult task rating, but an ability to complete the task. Progressing a task may include: changing the task, addition of resistance, increasing the range of motion required for task success, and increasing the duration of contraction. The number of total repetitions and activity outcomes will be recorded.
  Arms: Rapael glove with Sham dAIH; Rapael glove with dAIH

SUMMARY:
The overall objective of this project is to investigate the effectiveness of daily acute intermittent hypoxia therapy (dAIH), coupled with massed practice training, to improve upper-extremity function in individuals with chronic incomplete cervical SCI.

DETAILED DESCRIPTION:
Specific Aim 1: Evaluate the effectiveness of a combined intervention utilizing dAIH and massed practice upper extremity training on arm and hand function in individuals with incomplete tetraplegia.

Specific Aim 2: Evaluate the effectiveness of a combined intervention utilizing dAIH therapy and robotic rehabilitation device-administered upper-extremity training on arm and hand function in persons with incomplete tetraplegia.

ELIGIBILITY:
Inclusion:

1. History of a non-progressive spinal cord injury, at or below C2, and at or above T1.
2. Between the ages of 18 - 75 years.
3. Time since injury must be at least 6 months if the injury was traumatic in nature. If the spinal cord injury is non-traumatic, participants must meet at least the initial 6-month criteria in addition to either no regression in symptoms for at least two years, per self-report or per medical monitor discretion.
4. Demonstrate voluntary motor activation in hand muscles, with a score of at least a 2 on at least one of the Prehension Ability grasp patterns of the GRASSP assessment (cylindrical grasp, lateral key pinch, and tip to tip pinch), on at least one upper extremity.
5. Ability to understand and the willingness to sign an informed consent.
6. At least a 10% change in isometric elbow strength above baseline, after a single bout of Acute Intermittent Hypoxia (AIH), during screening.

Exclusion:

1. Diagnosed with any of the following medical conditions: congestive heart failure, cardiac arrhythmias, uncontrolled hypertension, uncontrolled diabetes mellitus, chronic obstructive pulmonary disease, emphysema, severe asthma, previous myocardial infraction, or known carotid/intracerebral artery stenosis.
2. Women who are currently pregnant/nursing or planning on becoming pregnant.
3. Individuals with a tracheostomy or who utilize mechanical ventilation.
4. Individuals who are currently enrolled in another interventional research study or in therapy related to upper extremity function.
5. Participants will be excluded if they have had a botulinum toxin injection to upper extremity musculature within the last 3 months. Participants will need to refrain from upper extremity botulinum toxin injections for the duration of the study. If participants wean off antispasticity medications to successfully complete the responsiveness to AIH screening session, they will need to refrain from the medications for the duration of the study.
6. Documented sleep apnea.
7. Orthopedic injuries or surgeries that would impact an individual's ability to use the upper extremity.
8. Traumatic brain injury or other neurological conditions that would impact the study.
9. Blood hemoglobin levels less than 10g/dL.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
GRASSP | up to 3 months
  The Graded Redefined Assessment of Strength, Sensibility and Prehension (GRASSP) is an extensive and validated impairment and functional measure which is able to detect subtle neurologic changes in individuals with spinal cord injury.
  Specifically, it evaluates the domains of sensation, strength, quality of different grip patterns and the ability to complete a variety of functional tasks.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Edward Hines, Jr. VA Hospital, Chicago, Illinois
  - Shirley Ryan AbilityLab, Chicago, Illinois
  - Kessler Foundation, East Hanover, New Jersey

IPD SHARING:
Plan to Share IPD: Undecided